CLINICAL TRIAL: NCT06845579
Title: Prediction of Blood Pressure Outcomes Following Renal Denervation (PREDICT-RDN)
Acronym: PREDICT-RDN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heart Center Leipzig - University Hospital (Other)
Collaborators: Helios Health Institute GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0108
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Uncontrolled Arterial Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renal sympathetic denervation (Other): All procedures will be carried out by highly experienced interventional cardiologists, each having performed a minimum of 20 RDN prior to treating study patients. All interventions will be performed with the CE-marked Symplicity SpyralTM (Medtronic, Minneapolis, MN, USA) renal denervation system following current treatment standards. Procedures will be performed as stated in the IFU. The specific ablation points will be determined by the discretion of the interventionalist.
  Interventions: Procedure: Renal sympathetic denervation

INTERVENTIONS:
Procedure: Renal sympathetic denervation — All procedures will be carried out by highly experienced interventional cardiologists, each having performed a minimum of 20 RDN prior to treating study patients. All interventions will be performed with the CE-marked Symplicity SpyralTM (Medtronic, Minneapolis, MN, USA) renal denervation system following current treatment standards. Procedures will be performed as stated in the IFU. The specific ablation points will be determined by the discretion of the interventionalist.

SUMMARY:
Prospective, single arm trial to assess the effects of renal denervation on day-by-day blood pressure measurements and time in blood pressure target range, as well as establish a multivariate prediction model for blood pressure reduction after renal denervation.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed arterial hypertension with systolic or diastolic blood pressure >140/90 mmHg in standardized office blood pressure measurement
2. Treatment with 3 to ≤5 antihypertensive drug classes
3. Age >18 years
4. Written informed consent

Exclusion Criteria:

1. Age ≤ 18 years
2. anatomy unsuitable for renal denervation (i.e. renal artery stenosis, single functioning kidney)
3. pregnancy
4. patients under legal supervision or guardianship
5. participation in other trials that might interfere with the study outcome according to the opinion of one of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | target range between months 4 to 6 (before renal denervation) vs. 10 to 12 (4 to 6 months after renal denervation)
  Difference in time in blood pressure target range between months 4 to 6 (before renal denervation) vs. 10 to 12 (4 to 6 months after renal denervation)

SECONDARY OUTCOMES:
Secondary endpoints | months 7 to 9
  Time in target range months 7 to 9
Secondary endpoints | one week before renal denervation vs. 6 months after renal denervation
  Change in conventional home blood pressure one week before renal denervation vs. 6 months after renal denervation
Secondary endpoints | up to 12 months
  Change in systemic sympathetic activity

CONTACTS AND LOCATIONS:
Overall Officials: Karl Fengler, Dr. med., Principal Investigator — Heart Center Leipzig
Locations (2):
- Germany (2):
  - Universitätsmedizin Mainz Kardiologie I, Mainz, Rheinland Pflanz
  - Heart Center Leipzig, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: No